CLINICAL TRIAL: NCT00511186
Title: A Phase-IIa, Double-blind, Randomized, Placebo-controlled Study on the Safety and Early Efficacy of Alkaline Phosphatase in Sepsis Patients With Renal Failure
Brief Title: A Study in Sepsis Patients With Renal Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: sufficient POC to switch development from bovine AP to recombinant AP
Sponsor: AM-Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AP REN 01-01
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Sepsis; Bacterial Infections and Mycoses
Keywords: Sepsis; Alkaline Phosphatase; inflammation; infection; renal failure
MeSH Terms: conditions — Sepsis; Bacterial Infections and Mycoses; Inflammation; Infections; Renal Insufficiency | interventions — 2-(3',4'-dihydroxyphenyl-1-azo)benzimidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bovine Intestinal AP (Experimental): Bovine Intestinal Alkaline Phosphatase (BIAP) Intravenous administration of 10" bolus (67,5U/kg) and 48h continuous infusion (132,5U/kg)
  Interventions: Drug: BIAP
- 2 (Placebo Comparator): Placebo Intravenous administration of 10" bolus and 48h continuous infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — placebo is administered intravenously over 48 hours. An initial loading dose of over 10-minutes is followed by continuous infusion over 48h.
  Arms: 2
Drug: BIAP — AP is administered intravenously over 48 hours. An initial loading dose of 67.5U/Kg body weight over 10-minutes is followed by continuous infusion of 132.5U/Kg/24H administered over 48H
  Other Names: AP
  Arms: Bovine Intestinal AP

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of AP in sepsis patients with renal failure and to investigate the effect of AP on inflammatory and clinical parameters in sepsis patients with renal failure.

DETAILED DESCRIPTION:
RATIONALE FOR THE STUDY

A previous clinical study conducted in centers in The Netherlands and Belgium have shown a substantial clinical benefit of AP treatment in patients with sepsis and associated acute renal failure (see Introduction above). The latter results require confirmation in a prospective study, as the current subject of this Protocol.

Choice of Drugs

The proposed study medication (AP) is identical to the study medication used in the previous clinical study in sepsis patients with single or multiple end-organ failure. Since there is no current proven treatment for these patients, the controls (as in previous studies) is placebo.

Choice of patient population

The aim is to enroll a maximum of 26 patients positive for sepsis with an APACHE score of ≥20 and ≤28 (determined within 24 hours of entry), and who will be analyzed on an intention to treat (ITT) basis.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the age of 18 and 80 years.
* Proven or suspected infection.
* Two out of four SIRS criteria of systemic inflammation, existing for less than 24 hours after admission in the intensive care unit, as follows:

  * Core temperature higher then 38 degree Celsius or lower then 36 degree Celsius.
  * Heart rate above 90 beats/min (unless the patient has a medical condition known to increase heart rate or is receiving treatment that would prevent tachycardia).
  * Respiratory rate above 20 breaths/min, a PaCO2 lower then 32mmHg or the use of mechanical ventilation for an acute respiratory process.
  * White-cell count above 12,000/mm3 or below 4,000/mm3 or a differential count showing >10 percent immature neutrophils.
* Acute renal failure, defined as

  * Rise in serum creatinine level to ≥150μmol/L within the previous 48 hours, in the absence of primary underlying renal disease OR
  * Minimally a stage 1 Kidney Injury according to AKIN creatinine criteria: Increase in serum creatinine ≥26.2µmol/L (0.3mg/dL) or increase to ≥150% (≥1.5 -fold) from baseline in the previous 48 hours in the absence of primary underlying renal disease and where baseline creatinine is less than 150 µmol/L) OR
  * Minimally a stage 1 Kidney Injury according to AKIN Urine Output criteria: Urine Output of ≤ 0.5mg/kg/h for ≥6h and following adequate fluid resuscitation when applicable, in the absence of underlying primary renal disease and where baseline creatinine is less than 150µmol/L)
* Written informed consent obtained prior to any study intervention.

Exclusion Criteria:

* Pregnant women or nursing mothers and fecund females who are not on effective contraception (chemical: pill; or mechanical: IUD)
* Patients already on dialysis (RTT) at entry
* Known HIV (sero-positive) patients
* Patients receiving immunosuppressant therapy or on chronic high doses of steroids equivalent to prednisone 1mg/Kg/day
* Patients expected to have rapidly fatal disease within 24 hours
* Known confirmed gram-positive sepsis
* Known confirmed fungal sepsis
* Acute pancreatitis with no established source of infection
* Patients not expected to survive for 28 days due to other medical conditions such as end-stage neoplasm or other diseases
* Participation in another investigational study within 90 days prior to start of the study which might interfere with this study
* Any previous administration of active study medication.
* Known allergy for dairy (bovine) products including cow milk.
* Sepsis without renal failure as defined in the Entry Criteria.
* History of chronic renal failure or history of persistent creatinine level equal or greater than 150umol/L prior to entry for reasons other than the current sepsis condition".

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Haematology, biochemistry, and microbiological evaluation. Adverse event monitoring. | 28 Days

SECONDARY OUTCOMES:
To investigate the effect of AP on inflammatory parameters in sepsis patients with renal failure. | 28 Days
To investigate the effect of AP on clinical variables in sepsis patients with renal failure. | 28 Days
To investigate the effect of AP on renal function markers in sepsis patients with renal failure. | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Professor J G van der Hoeven, MD, PhD, Principal Investigator — University Medical Center St Radboud, Nijmegen, The Netherlands
Locations (9):
- Belgium (4):
  - University Medical Center Antwerp (UZA), Antwerp
  - Cliniques Universitaires Saint Luc-UCL, Brussels
  - ULB Hopital Erasme, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
- Netherlands (5):
  - UMC Nijmegen University Medical Center St Radboud, Nijmegen, Gelderland
  - Isala Clinics, Zwolle, Overijssel
  - Jeroen Bosch Ziekenhuis lokatie GZG, 's-Hertogenbosch
  - VU University Medical Center, Amsterdam
  - Canisius Wilhelmina Ziekenhuis, Nijmegen

REFERENCES:
- [Result] Pickkers P, Heemskerk S, Schouten J, Laterre PF, Vincent JL, Beishuizen A, Jorens PG, Spapen H, Bulitta M, Peters WH, van der Hoeven JG. Alkaline phosphatase for treatment of sepsis-induced acute kidney injury: a prospective randomized double-blind placebo-controlled trial. Crit Care. 2012 Jan 23;16(1):R14. doi: 10.1186/cc11159. PMID 22269279
- See also: Related Info — http://www.am-pharma.com